CLINICAL TRIAL: NCT01348737
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel-group Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect on Biomarkers of AZD3839 Including an Open-label Food Effect Group in Healthy Male and Female Volunteers of Non-childbearing Potential
Brief Title: Assessment of Safety, Tolerability and Blood Concentrations of Single Doses of AZD3839 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D4080C00001; 2011-001337-16
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Alzheimer's Disease; Safety; Tolerability; Blood Concentration; Healthy Volunteers
Keywords: Phase 1; healthy volunteers; double-blind; placebo-controlled; AZD3839; pharmacokinetics; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — AZD3839

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- AZD3839 (Experimental): Oral Treatment
  Interventions: Drug: AZD3839
- AZD3839 Placebo (Placebo Comparator): Oral Treatment
  Interventions: Drug: AZD3839 Placebo

INTERVENTIONS:
Drug: AZD3839 — Single Oral Dose
  Arms: AZD3839
Drug: AZD3839 Placebo — Single Oral Dose
  Arms: AZD3839 Placebo

SUMMARY:
The purpose of the study is to assess the safety, tolerability and blood concentration of AZD3839 following oral administration of single doses in healthy men and women of non-childbearing potential

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers of non-childbearing potential aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 (inclusive) and weigh between 50 kg and 100 kg (inclusive)
* Creatinine clearance in the normal range (>80 mL/min estimated according to Cockroft-Gault)
* Healthy volunteers should have a serum potassium concentration of ≥3.8 mmol/L at screening (Visit 1) and on admission to the study centre (Day -1)
* Clinically normal findings on physical examination in relation to age, as judged by the Investigator

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the results or the healthy volunteer's ability to participate in the study
* History of psychotic disorder amongst first degree relatives
* Significant orthostatic reaction at enrolment as judged by the Investigator
* Prolonged QTcF greater than 450 msec or shortened QTcF less than 340 msec or family history of long QT syndrome or sudden death
* Healthy volunteer is a vegetarian/lactose intolerant (exclusion criterion only applicable for healthy volunteers participating in Part 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Event as a measure of safety and tolerability of AZD3839 (Part 1) | Part 1 - AEs will be collected from admission to the study centre (Visit 2, Day-1) until the follow-up visit (Visit 3) approximately 15 days
Number of Adverse Events as a measure of Safety and tolerability of AZD3839 (Part 2) | Part 2 - AEs will be collected from admission to the study centre (Visit 2, Day-1) until the follow-up visit (Visit 4) approximately 20 days

SECONDARY OUTCOMES:
Time at which maximum concentration occurs in AZD3839 (Part 1) | pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours after the administration of the investigational product, as well as on Day 4 and at the follow-up visit (Visit 3)
Maximum observed concentration of AZD3839 in plasma (Part 1) | Part 1 - pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours after the administration of the investigational product, as well as on Day 4 and at the follow-up visit (Visit 3)
Time at which maximum concentration occurs in AZD3839 (Part 2) | Part 2 - at pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours after the Administration. May be taken at the follow-up visit (Visit 4)
Maximum observed concentration of AZD3839 in plasma (Part 2) | Part 2 - at pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Dr Darren Wilbraham, MBBS DCPSA, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Dr Paul Bjornsson, Study Director — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom